CLINICAL TRIAL: NCT05370170
Title: Effect of Implementing Ottawa Nutritional Guidelines on the Course of Nausea and Vomiting During Pregnancy (A Randomized Control Trial)
Brief Title: Ottawa Nutritional Guidelines for Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noura Mohamed Eltoukhy, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IORG0003381
Record Dates: First submitted 2022-03-30; First posted 2022-05-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Nausea Gravidarum
MeSH Terms: interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine antenatal care (No Intervention): the control group will receive routine antenatal care and will not receive the guidelines group included 30 cases
- Ottawa guidelines (Experimental): study group will receive routine antenatal care in addition to the Ottawa nutritional guidelines group included 30 cases
  Interventions: Behavioral: Acupressure and nutritional advices

INTERVENTIONS:
Behavioral: Acupressure and nutritional advices — Teaching using booklets and application of acupressure
  Arms: Ottawa guidelines

SUMMARY:
Effect of Implementing Ottawa Nutritional Guidelines on the Course of Nausea and Vomiting During Pregnancy (A Randomized Control Trial)

DETAILED DESCRIPTION:
Studying the Effect of Implementing Ottawa Nutritional Guidelines on the Course of Nausea and Vomiting During Pregnancy (A Randomized Control Trial) using no pharmacological agents and life style modification in addition to acupressure to treat nausea and vomiting of pregnancy

ELIGIBILITY:
Inclusion Criteria:

1. primigravida
2. gestational age of 7-13 weeks
3. singleton pregnancy
4. having a score of 7-12 on the (PUQE 24)
5. can read and write
6. having phone number
7. not receiving medications for reducing NVP, except for vitamin B6
8. wanted pregnancy.

Exclusion Criteria:

1. subject's unwillingness to continue the study
2. occurrence of obstetric complications during the study
3. hyper-emesis gravidarum
4. having physical or mental disorders
5. having oral/speech impairments
6. having assisted reproductive techniques for the present pregnancy
7. having two consecutive miscarriages before the current pregnancy
8. old primigravida
9. narcotic use or alcohol drinking
10. and subjects who will show signs and symptoms of hyperemesis gravidarum during the study will be dropped out and referred to medical care.

Ages: 22 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
control nausea and vomiting | 3 weeks
  control the frequency and severity of nausea and vomiting and measure it by using Pregnancy Unique Quantification of Emesis

SECONDARY OUTCOMES:
maintain normal body weight and prevent hospitalization | 3 weeks
  Monitor mother weight by calipered weight scale to monitor weight loss related to nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Noura Mo Eltoukhi, PhD, Principal Investigator — Cairo University; Noura M Eltoukhi, lecturer, Principal Investigator — Faculty of Nursing Cairo University
Locations (1):
- Faculty of Nursing, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with researchers upon reasonable request following publication of the main results."
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: "IPD will be available starting after publication and will remain available
Access Criteria: Access to the de-identified individual participant data will be granted to qualified researchers with a methodologically sound proposal. Requests should be submitted to the study sponsor or principal investigator and will be reviewed by a data access committee

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-10-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT05370170/Prot_SAP_ICF_000.pdf